CLINICAL TRIAL: NCT01000974
Title: Phase III, Partially Double-blind Study to Evaluate Consistency and Immunogenicity of 3 Lots of GSK Biologicals' Hib Conjugate Vaccine 208108 Versus ActHIB and Pentacel at 2, 4, 6 and 15-18 Months of Age in Healthy Infants
Brief Title: Consistency & Immunogenicity Study of 3 Lots of GSK's Hib Conjugate Vaccine Versus ActHIB & Pentacel in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112957
Record Dates: First submitted 2009-10-22; First posted 2009-10-23 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Haemophilus Influenzae Type b
Keywords: primary vaccination course; Haemophilus influenzae type b; infants, children; booster vaccination; immunogenicity; safety; Gram-negative bacterial infections; vaccines, conjugate
MeSH Terms: conditions — Haemophilus Infections; Gram-Negative Bacterial Infections | interventions — Hiberix; Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; pentacel; PEDIARIX; 13-valent pneumococcal vaccine; RIX4414 vaccine; Diphtheria-Tetanus-acellular Pertussis Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Hiberix Group (Experimental): Pooled group of subjects, male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination, who received 3 doses of 3 different lots of Hiberix® vaccine co-administered with 3 doses of Pediarix® and Prevnar13® vaccines at 2, 4 and 6 months of age and 2 doses of Rotarix® vaccine at 2 and 4 months of age The Hiberix® vaccine was administered intramuscularly in the right thigh. Pediarix® vaccine was administered intramuscularly in the left thigh. The Prevnar13® vaccine was administered intramuscularly in the left thigh or deltoid. The Rotarix® vaccine was administered orally.
  Interventions: Biological: GSK Biologicals' Haemophilus influenzae type b vaccine (GSK 208108); Biological: Pediarix™; Biological: Prevnar 13™; Biological: Rotarix™; Biological: Infanrix™
- ActHIB Group (Active Comparator): Subjects, male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination, who received 3 doses of ActHIB® vaccine co-administered with 3 doses of Pediarix® and Prevnar13® vaccines at 2, 4 and 6 months of age and 2 doses of Rotarix® vaccine at 2 and 4 months of age. The ActHIB® vaccine was administered intramuscularly in the right thigh. The Pediarix® vaccine was administered intramuscularly in the left thigh. The Prevnar13® vaccine was administered intramuscularly in the left thigh or deltoid. The Rotarix® vaccine was administered orally.
  Interventions: Biological: ActHIB™; Biological: Pediarix™; Biological: Prevnar 13™; Biological: Rotarix™; Biological: Infanrix™
- Pentacel Group (Active Comparator): Subjects, male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination, who received 3 doses of Pentacel® vaccine co-administered with 3 doses of Prevnar13® vaccine, 2 or 3 doses of Engerix™-B vaccine at 2, 4 and 6 months of age and 2 doses of Rotarix® vaccine at 2 and 4 months of age. The Pentacel® vaccine was administered intramuscularly in the right thigh. The Engerix™-B vaccine was administered intramuscularly in the left thigh. The Prevnar13® vaccine was administered intramuscularly in the left thigh or deltoid. The Rotarix® vaccine was administered orally. If subjects in the Pentacel Group had received a birth dose of Hepatitis B vaccine then they were to receive Engerix™-B vaccine only at 2 and 6 months of age.
  Interventions: Biological: Pentacel™; Biological: Prevnar 13™; Biological: Rotarix™; Biological: Engerix™-B

INTERVENTIONS:
Biological: GSK Biologicals' Haemophilus influenzae type b vaccine (GSK 208108) — Three doses of 3 different manufacturing lots in primary study at 2, 4 and 6 months of age as intramuscular injection and one dose as booster vaccination.
  Other Names: Hiberix®
  Arms: Hiberix Group
Biological: ActHIB™ — Three doses in primary epoch at 2, 4 and 6 months of age as intramuscular injection and one dose as a booster vaccination
  Arms: ActHIB Group
Biological: Pentacel™ — Three doses in primary epoch at 2, 4 and 6 months of age as intramuscular injection and one dose as a booster vaccination
  Arms: Pentacel Group
Biological: Pediarix™ — Three doses in primary epoch at 2, 4 and 6 months of age as intramuscular injection
  Arms: ActHIB Group; Hiberix Group
Biological: Prevnar 13™ — Three doses in primary epoch at 2, 4 and 6 months of age as intramuscular injection
Biological: Rotarix™ — Two oral doses in primary epoch at 2 and 4 months of age
Biological: Engerix™-B — Two or three doses in primary epoch at 2,( 4) and 6 months of age as intramuscular injection
  Arms: Pentacel Group
Biological: Infanrix™ — One dose in the booster epoch at 15-18 months of age as intramuscular injection
  Arms: ActHIB Group; Hiberix Group

SUMMARY:
The purpose of this study is to evaluate safety, to demonstrate lot-to-lot consistency of the vaccine, to address the relevant concomitant vaccine administrations and to provide a comparison between GSK Biologicals' Hib conjugate vaccine and the licensed monovalent Hib vaccine ActHIB as well as the licensed combination product Pentacel in infants at 2, 4, 6 and 15-18 months of age. This study is designed with a primary and a booster phase.

DETAILED DESCRIPTION:
This protocol posting has been updated following protocol amendment 3, dated 12 April 2011. The impacted section is: Eligibility Criteria (Exclusion criteria).

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR[s]) can and will comply with the requirements of the protocol (e.g., completion of the diary card, return for follow-up visits).
* A male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the subject's parent/LAR.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of minimum 36 weeks.
* Infants who have not received a previous dose of hepatitis B vaccine or those who have received only 1 dose of hepatitis B vaccine administered at least 30 days prior to enrollment.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of study vaccine and until 30 days after the booster dose.
* Previous vaccination against Haemophilus influenzae type b, diphtheria, tetanus, pertussis, Pneumococcus, rotavirus and/or poliovirus; more than one previous dose of hepatitis B vaccine.
* History of Haemophilus influenzae type b, diphtheria, tetanus, pertussis, pneumococcal, rotavirus, poliovirus, and hepatitis B diseases.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines, including dry natural latex rubber.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at time of enrollment. All vaccines can be administered to persons with a minor illness.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Concurrent participation in another clinical study, up to 30 days prior to study entry or at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Child in care.
* History of intussusception.
* History of uncorrected congenital malformation of the gastrointestinal tract that would predispose the infant to intussusception.
* History of Severe Combined Immunodeficiency Disease.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4003 (Actual)
Dates: Start 2010-06-18; Primary Completion 2011-11-18 (Actual); Study Completion 2013-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (62):
- United States (62):
  - GSK Investigational Site, Dothan, Alabama
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Fayetteville, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Antioch, California
  - GSK Investigational Site, Daly City, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fremont, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Hayward, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Redwood City, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Jose, California
  - GSK Investigational Site, Santa Clara, California
  - GSK Investigational Site, Santa Rosa, California
  - GSK Investigational Site, Vallejo, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Boulder, Colorado
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Orange City, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, Honolulu, Hawaii
  - GSK Investigational Site, Waipio, Hawaii
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Greenville, Pennsylvania
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Roy, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, South Jordan, Utah
  - GSK Investigational Site, Syracuse, Utah
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Marshfield, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Hiberix Group: Pooled group of subjects, male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination, who received 3 doses of 3 different lots of Hiberix vaccine co-administered with 3 doses of Pediarix and Prevnar13 vaccines at 2, 4 and 6 months of age and 2 doses of Rotarix vaccine at 2 and 4 months of age. The Hiberix vaccine was administered intramuscularly in the right thigh. Pediarix vaccine was administered intramuscularly in the left thigh. The Prevnar13 vaccine was administered intramuscularly in the left thigh or deltoid. The Rotarix vaccine was administered orally.
- ActHIB Group: Subjects, male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination, who received 3 doses of ActHIB vaccine co-administered with 3 doses of Pediarix and Prevnar13 vaccines at 2, 4 and 6 months of age and 2 doses of Rotarix vaccine at 2 and 4 months of age. The ActHIB vaccine was administered intramuscularly in the right thigh. The Pediarix vaccine was administered intramuscularly in the left thigh. The Prevnar13 vaccine was administered intramuscularly in the left thigh or deltoid. The Rotarix vaccine was administered orally.
- Pentacel Group: Subjects, male or female between, and including, 6 and 12 weeks of age at the time of the first vaccination, who received 3 doses of Pentacel vaccine co-administered with 3 doses of Prevnar13 vaccine, 2 or 3 doses of Engerix-B vaccine at 2, 4 and 6 months of age and 2 doses of Rotarix vaccine at 2 and 4 months of age. The Pentacel vaccine was administered intramuscularly in the right thigh. The Engerix-B vaccine was administered intramuscularly in the left thigh. The Prevnar13 vaccine was administered intramuscularly in the left thigh or deltoid. The Rotarix vaccine was administered orally. If subjects in the Pentacel Group had received a birth dose of Hepatitis B vaccine then they were to receive Engerix-B vaccine only at 2 and 6 months of age.
Period: Primary Vaccination Phase
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Started | 2963 | 520 | 520
Completed | 2625 | 470 | 457
Not Completed | 338 | 50 | 63
Not completed — Withdrawal by Subject | 109 | 17 | 21
Not completed — Lost to Follow-up | 171 | 19 | 26
Not completed — Protocol Violation | 40 | 3 | 2
Not completed — Adverse Event | 14 | 2 | 2
Not completed — Other | 4 | 9 | 12
Period: Booster Vaccination Phase
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Started | 2337 | 435 | 400
Completed | 2270 | 423 | 386
Not Completed | 67 | 12 | 14
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Lost to Follow-up | 40 | 5 | 7
Not completed — Other | 24 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group | Total
Number analyzed (Participants) | 2963 | 520 | 520 | 4003
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 8.6 (1.08) | 8.6 (1.13) | 8.7 (1.12) | 8.61 (1.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1424 | 271 | 258 | 1953
  Male | 1539 | 249 | 262 | 2050

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations Greater Than or Equal to (≥) 0.15 Microgram Per Milliliter (µg/mL) and ≥ 1.0 µg/mL
Description: Non-inferiority of Hiberix to ActHIB, each co-administered with Pediarix, Prevnar13 and Rotarix following 3 primary doses in terms of immune response to PRP (Anti-PRP≥ 0.15 µ g/ml and ≥1.0 µg/mL).
Time Frame: At 1 month after last dose of primary vaccination
Population: The analysis was based on the Primary According-to-Protocol (ATP) cohort for immunogenicity, including all evaluable subjects with 3 vaccine doses administered and assay results available for antibodies against at least one antigen for the blood sample taken 1 month after the last vaccine dose.
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 1590 | 274 | 253
Subjects
  Anti-PRP ≥ 0.15 µg/mL | 1536 | 265 | 234
  Anti-PRP ≥ 1.0 µg/mL | 1291 | 246 | 198
Statistical Analysis 1: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-PRP concentration ≥ 1.0 μg/mL; Test type: Non-Inferiority — To demonstrate the non-inferiority of Test Hib to Control Hib, each co-administered with DTPa-HBV-IPV, 13Pn and HRV vaccines, following 3 primary vaccine doses in terms of anti-PRP antibody concentration ≥ 1.0 μg/mL; Non-inferiority analysis; difference in percentage = -8.59, 95% CI 2-sided [-12.28 to -4.07]
Statistical Analysis 2: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-PRP concentration≥ 0.15 μg/mL; Test type: Non-Inferiority — To demonstrate the non-inferiority of Test Hib to Control Hib, each co-administered with DTPa-HBVIPV, 13Pn and HRV vaccines, following 3 primary vaccine doses in terms of anti-PRP antibody concentrations ≥ 0.15 μg/mL; Non-inferiority analysis; Difference in percentage = -0.11, 95% CI 2-sided [-1.98 to 2.82]

2. Primary Outcome: Number of Subjects With Anti-Protein-D (Anti-D) and Anti-Protein-T (Anti-T) Antibody Concentrations ≥ 0.1 International Units Per Milliliter (IU/mL)
Description: Non-inferiority of Pediarix co-administered with Hiberix, Prevnar13 and Rotarix compared to Pediarix co-administered with ActHIB, Prevnar13 and Rotarix following 3 primary vaccine doses in terms of immune response to Diphtheria, Tetanus.
Time Frame: At 1 month after last dose of primary vaccination
Population: The analysis was based on the Primary According-to-Protocol (ATP) cohort for immunogenicity, including all evaluable subjects with 3 vaccine doses administered and for whom assay results were available for antibodies against at least one antigen for the blood sample taken 1 month after the last vaccine dose.
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 393 | 274 | 250
Subjects
  Anti-D: number analyzed (Participants) | 393 | 273 | 250
  Anti-D | 393 | 273 | 249
  Anti-T | 393 | 274 | 249
Statistical Analysis 1: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-D antibody concentrations; Test type: Non-Inferiority — To demonstrate the non-inferiority of DTPa-HBV-IPV co-administered with Test Hib, 13Pn and HRV to DTPa-HBV-IPV co-administered with Control Hib, 13Pn and HRV, following 3 primary vaccine doses in terms of immune response to diphtheria (Anti-D); Non-inferiority analysis; Difference in percentage = 0, 95% CI 2-sided [-1.26 to 1.81]
Statistical Analysis 2: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-T antibody concentrations; Test type: Non-Inferiority — To demonstrate the non-inferiority of DTPa-HBV-IPV co-administered with Test Hib, 13Pn and HRV to DTPa-HBV-IPV co-administered with Control Hib, 13Pn and HRV, following 3 primary vaccine doses in terms of immune response to tetanus (Anti-T); Non-inferiority analysis; Difference in percentage = 0, 95% CI 2-sided [-1.26 to 1.8]

3. Primary Outcome: Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations
Description: Antibody concentrations were given as Geometric Mean Concentrations (GMCs) expressed in micrograms per milliliter (µg/mL).
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 1590 | 274 | 253
µg/mL | 5.193 [4.765 to 5.658] | 6.743 [5.593 to 8.129] | 3.640 [2.891 to 4.583]

4. Primary Outcome: Anti-pertussis Toxoid (Anti-PT), Anti-pertactin (Anti-PRN) and Anti-filamentous Hemagglutinin (Anti-FHA) Antibody Concentrations
Description: Antibody concentrations were given as geometric mean concentrations (GMCs) expressed as enzyme-linked immuno-sorbent assay (ELISA) units per milliliter i.e. EL.U/mL.
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 792 | 275 | 251
EL.U/mL
  Anti-PT | 73.2 [69.8 to 76.6] | 71.9 [66.6 to 77.6] | 41.9 [38.4 to 45.8]
  Anti-PRN: number analyzed (Participants) | 789 | 275 | 250
  Anti-PRN | 111.6 [104.5 to 119.2] | 93.5 [83.7 to 104.4] | 51.9 [45.4 to 59.3]
  Anti-FHA: number analyzed (Participants) | 791 | 275 | 249
  Anti-FHA | 321.8 [307.0 to 337.3] | 295.8 [276.0 to 317.0] | 174.8 [160.0 to 191.0]
Statistical Analysis 1: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority GMC ratio anti-PT; Test type: Non-Inferiority — To demonstrate the non-inferiority of DTPa-HBV-IPV co-administered with Test Hib, 13Pn and HRV to DTPa-HBV-IPV co-administered with Control Hib, 13Pn and HRV, following 3 primary vaccine doses in terms of immune response to pertussis toxoid [PT]; Non-inferiority analysis; GMC ratio = 1.017, 97.5% CI 2-sided [0.918 to 1.127]
Statistical Analysis 2: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority GMC ratio anti-FHA; Test type: Non-Inferiority — To demonstrate the non-inferiority of DTPa-HBV-IPV co-administered with Test Hib, 13Pn and HRV to DTPa-HBV-IPV co-administered with Control Hib, 13Pn and HRV, following 3 primary vaccine doses in terms of immune response to filamentous hemagglutinin [FHA]; Non-inferiority analysis; GMC ratio = 1.088, 97.5% CI 2-sided [0.983 to 1.204]
Statistical Analysis 3: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority GMC ratio anti-PRN; Test type: Non-Inferiority — To demonstrate the non-inferiority of DTPa-HBV-IPV co-administered with Test Hib, 13Pn and HRV to DTPa-HBV-IPV co-administered with Control Hib, 13Pn and HRV, following 3 primary vaccine doses in terms of immune response to pertactin [PRN]; Non-inferiority analysis; GMC ratio = 1.193, 97.5% CI 2-sided [1.03 to 1.382]

5. Primary Outcome: Anti-Streptococcus Pneumoniae (S.Pneumoniae) Antibody Concentrations
Description: Antibody concentrations against S.pneumoniae were given as geometric mean concentrations (GMCs) expressed as microgram per milliliter (µg/mL).
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 389 | 270 | 247
µg/mL
  Anti-Pneumoniae 1: number analyzed (Participants) | 384 | 268 | 245
  Anti-Pneumoniae 1 | 2.515 [2.318 to 2.729] | 2.500 [2.278 to 2.745] | 2.442 [2.190 to 2.722]
  Anti-Pneumoniae 3: number analyzed (Participants) | 382 | 269 | 245
  Anti-Pneumoniae 3 | 1.056 [0.976 to 1.142] | 1.008 [0.933 to 1.089] | 1.190 [1.066 to 1.329]
  Anti-Pneumoniae 4: number analyzed (Participants) | 389 | 268 | 247
  Anti-Pneumoniae 4 | 1.804 [1.684 to 1.932] | 1.803 [1.662 to 1.957] | 1.819 [1.645 to 2.011]
  Anti-Pneumoniae 5: number analyzed (Participants) | 379 | 266 | 246
  Anti-Pneumoniae 5 | 3.729 [3.409 to 4.079] | 3.656 [3.308 to 4.040] | 3.530 [3.128 to 3.984]
  Anti-Pneumoniae 6A: number analyzed (Participants) | 381 | 267 | 244
  Anti-Pneumoniae 6A | 3.442 [3.177 to 3.729] | 3.340 [3.032 to 3.679] | 3.384 [3.046 to 3.760]
  Anti-Pneumoniae 6B: number analyzed (Participants) | 383 | 267 | 245
  Anti-Pneumoniae 6B | 1.065 [0.950 to 1.196] | 0.994 [0.860 to 1.148] | 0.875 [0.757 to 1.013]
  Anti-Pneumoniae 7F: number analyzed (Participants) | 386 | 269 | 246
  Anti-Pneumoniae 7F | 4.518 [4.192 to 4.870] | 4.115 [3.777 to 4.484] | 3.785 [3.412 to 4.199]
  Anti-Pneumoniae 9V: number analyzed (Participants) | 386 | 270 | 246
  Anti-Pneumoniae 9V | 2.516 [2.305 to 2.746] | 2.431 [2.204 to 2.681] | 2.226 [1.976 to 2.507]
  Anti-Pneumoniae 14: number analyzed (Participants) | 384 | 267 | 244
  Anti-Pneumoniae 14 | 4.506 [4.105 to 4.946] | 4.111 [3.672 to 4.602] | 3.938 [3.472 to 4.466]
  Anti-Pneumoniae 18C: number analyzed (Participants) | 380 | 267 | 244
  Anti-Pneumoniae 18C | 3.655 [3.351 to 3.986] | 3.507 [3.196 to 3.848] | 3.401 [3.033 to 3.814]
  Anti-Pneumoniae 19A: number analyzed (Participants) | 384 | 266 | 245
  Anti-Pneumoniae 19A | 1.556 [1.433 to 1.689] | 1.553 [1.391 to 1.735] | 1.321 [1.175 to 1.486]
  Anti-Pneumoniae 19F: number analyzed (Participants) | 384 | 268 | 245
  Anti-Pneumoniae 19F | 2.745 [2.552 to 2.952] | 2.833 [2.613 to 3.072] | 2.531 [2.315 to 2.766]
  Anti-Pneumoniae 23F: number analyzed (Participants) | 384 | 268 | 245
  Anti-Pneumoniae 23F | 2.046 [1.846 to 2.267] | 1.985 [1.765 to 2.232] | 1.670 [1.444 to 1.931]
Statistical Analysis 1: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 1 concentrations; Test type: Non-Inferiority — To demonstrate the non-inferiority of a 3-dose primary vaccination course of 13Pn co-administered with Test Hib, HRV and DTPa-HBV-IPV compared to that of 13Pn co-administered with Control Hib, HRV and DTPa-HBV-IPV in terms of Streptococcus pneumoniae (S.pneumoniae) GMCs; Non-inferiority analysis; GMC ratio = 1.006, 97.5% CI 2-sided [0.873 to 1.159]
Statistical Analysis 2: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 3 concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.048, 97.5% CI 2-sided [0.921 to 1.192]
Statistical Analysis 3: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 4 concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.001, 97.5% CI 2-sided [0.886 to 1.13]
Statistical Analysis 4: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 5 concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.02, 97.5% CI 2-sided [0.874 to 1.19]
Statistical Analysis 5: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 6A concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.031, 97.5% CI 2-sided [0.894 to 1.188]
Statistical Analysis 6: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 6B concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.072, 97.5% CI 2-sided [0.871 to 1.32]
Statistical Analysis 7: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 7F concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.098, 97.5% CI 2-sided [0.964 to 1.251]
Statistical Analysis 8: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 9V concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.035, 97.5% CI 2-sided [0.89 to 1.204]
Statistical Analysis 9: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 14 concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.096, 97.5% CI 2-sided [0.929 to 1.294]
Statistical Analysis 10: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 18C concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.042, 97.5% CI 2-sided [0.9 to 1.207]
Statistical Analysis 11: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 19A concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.001, 97.5% CI 2-sided [0.859 to 1.167]
Statistical Analysis 12: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 19F concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 0.969, 97.5% CI 2-sided [0.855 to 1.098]
Statistical Analysis 13: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Pneumoniae 23F concentrations; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Non-inferiority analysis; GMC ratio = 1.031, 97.5% CI 2-sided [0.862 to 1.232]

6. Primary Outcome: Number of Subjects With Seroresponse (95%) to Anti-pertussis Toxoid (Anti-PT), Anti-pertactin (Anti-PRN) and Anti-filamentous Hemagglutinin (Anti-FHA)
Description: Seroresponse (95%) was defined as the number of subjects showing a concentration above a threshold that leads to 95% seroresponse in the ActHIB group.
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 792 | 275 | 251
Subjects
  Anti-PT | 764 | 264 | 201
  Anti-PRN: number analyzed (Participants) | 789 | 275 | 250
  Anti-PRN | 762 | 262 | 213
  Anti-FHA: number analyzed (Participants) | 791 | 275 | 249
  Anti-FHA | 744 | 263 | 191
Statistical Analysis 1: Comparison: Hiberix Group vs ActHIB Group; Difference in seroresponse Anti-FHA; Test type: Other — To rule out 10% decrease in seroresponse to FHA in subjects receiving DTPa-HBV-IPV coadministered with Test Hib,13Pn & HRV vaccines compared to subjects receiving DTPa-HBV-IPV co-administered with Control Hib, 13Pn &HRV vaccines,following 3 primary vaccine doses where seroresponse wasdefined as percentage of subjects showing aconcentration above a threshold that led to 95% seroresponse in control; p < 0.0001, t-test, 1 sided; P-value is computed by integrating on the p-values of one-sided test with alpha=0.025 & the posterior probability of the cut-off in the control group
Statistical Analysis 2: Comparison: Hiberix Group vs ActHIB Group; Difference in seroresponse Anti-PT; Test type: Other — To rule out 10% decrease in seroresponse to PT in subjects receiving DTPa-HBV-IPV coadministered with Test Hib,13Pn & HRV vaccines compared to subjects receiving DTPa-HBV-IPV co-administered with Control Hib, 13Pn &HRV vaccines,following 3 primary vaccine doses where seroresponse wasdefined as percentage of subjects showing aconcentration above a threshold that led to 95% seroresponse in control; p < 0.0001, t-test, 1 sided — P-value is computed by integrating on the p-values of one-sided test with alpha=0.025 and the posterior probability of the cut-off in the control group
Statistical Analysis 3: Comparison: Hiberix Group vs ActHIB Group; Difference in seroresponse Anti-PRN; Test type: Other — To rule out 10% decrease in seroresponse to PRN in subjects receiving DTPa-HBV-IPV coadministered with Test Hib,13Pn & HRV vaccines compared to subjects receiving DTPa-HBV-IPV co-administered with Control Hib, 13Pn &HRV vaccines,following 3 primary vaccine doses where seroresponse wasdefined as percentage of subjects showing aconcentration above a threshold that led to 95% seroresponse in control; p < 0.0001, t-test, 1 sided — [p-value comment as in outcome 6, analysis 2]

7. Primary Outcome: Number of Subjects With Anti-Polio 1,2,3 Antibody Titres Greater Than or Equal to Cut-off Value
Description: The cut-off value was defined as a concentration ≥ 8 ED50 (ED50 is the concentration at which the protein exhibits 50% of its maximum activity).
  The polio testing which started at the Biomnis laboratory was stopped because the polio virus micro-neutralization assays were found to be not in line with the quality standards defined in GSK Biologicals' SOPs. As a result, polio testing was restarted at the GSK laboratory and the results were uploaded into the clinical database.
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 280 | 192 | 189
Subjects
  Anti-Polio 1: number analyzed (Participants) | 248 | 181 | 175
  Anti-Polio 1 | 246 | 181 | 164
  Anti-Polio 2 | 275 | 188 | 183
  Anti-Polio 3: number analyzed (Participants) | 257 | 181 | 169
  Anti-Polio 3 | 254 | 181 | 168
Statistical Analysis 1: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Polio 1 concentrations; Test type: Non-Inferiority — To demonstrate the non-inferiority of DTPa-HBV-IPV co-administered with Test Hib, 13Pn and HRV to DTPa-HBV-IPV co-administered with Control Hib, 13Pn and HRV, following 3 primary vaccine doses in terms of immune response to poliovirus 1; Non-inferiority analysis; Difference in percentage = -0.67, 97.5% CI 2-sided [-2.24 to 0.87]
Statistical Analysis 2: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Polio 2 concentration; Test type: Non-Inferiority — To demonstrate the non-inferiority of DTPa-HBV-IPV co-administered with Test Hib, 13Pn and HRV to DTPa-HBV-IPV co-administered with Control Hib, 13Pn and HRV, following 3 primary vaccine doses in terms of immune response to poliovirus 2; Non-inferiority analysis; Difference in percentage = 0.45, 97.5% CI 2-sided [-1.45 to 2.91]
Statistical Analysis 3: Comparison: Hiberix Group vs ActHIB Group; Non-inferiority Anti-Polio 3 concentration; Test type: Non-Inferiority — To demonstrate the non-inferiority of DTPa-HBV-IPV co-administered with Test Hib, 13Pn and HRV to DTPa-HBV-IPV co-administered with Control Hib, 13Pn and HRV, following 3 primary vaccine doses in terms of immune response to poliovirus 3; Non-inferiority analysis; Difference in percentage = -0.66, 97.5% CI 2-sided [-2.2 to 0.88]

8. Primary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations ≥ 1.0 µg/mL
Description: Non-inferiority of a booster dose of Hiberix co-administered with Infanrix in subjects 15-18 months of age who received 3 primary vaccine doses of Hiberix to a booster dose of ActHIB co-administered with Infanrix in subjects of 15-18 months of age who received 3 primary vaccine doses of ActHIB in terms of immune response to PRP
Time Frame: At 1 month after booster vaccination
Population: The analysis was performed on the Booster According-to-Protocol (ATP) cohort for immunogenicity that included all evaluable subjects for whom assay results were available for antibodies against at least 1 antigen for the blood sample taken 1 month after the administration of the booster vaccine dose
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 336 | 236 | 186
Subjects | 333 | 231 | 184

9. Secondary Outcome: Anti-protein-D (Anti-D) and Anti-protein-T (Anti-T) Antibody Concentrations
Description: Antibody concentrations were given as geometric mean concentrations (GMCs) and expressed as International Units per milliliter (IU/mL).
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 393 | 274 | 250
IU/mL
  Anti-D: number analyzed (Participants) | 393 | 273 | 250
  Anti-D | 2.72 [2.54 to 2.93] | 2.45 [2.24 to 2.68] | 1.88 [1.69 to 2.09]
  Anti-T | 2.23 [2.07 to 2.41] | 2.44 [2.20 to 2.71] | 1.72 [1.55 to 1.91]

10. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any symptom regardless of intensity grade.
Time Frame: During a 4-day follow-up period (Days 0-3) following any vaccination
Population: The analysis was based on the Primary Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine dose documented and with symptom sheets completed.
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2846 | 503 | 496
Subjects
  Any pain | 1932 | 366 | 370
  Any redness | 1165 | 233 | 257
  Any swelling | 834 | 174 | 195

11. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, fever and loss of appetite. Any = occurrence of any general symptom regardless of intensity grade or relationship to vaccination. Any fever= Rectal temperature equal to or above (≥) 38 degrees Celsius (°C).
Time Frame: During a 4-day follow-up period (Days 0-3) following any vaccination
Population: The analysis was based on the Primary Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine dose documented and symptom sheets completed.
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2848 | 503 | 496
Subjects
  Any drowsiness | 2179 | 398 | 378
  Any irritability | 2478 | 449 | 434
  Any loss of appetite | 1450 | 275 | 253
  Any fever | 1014 | 186 | 143

12. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Day 0-Day 30) follow-up period after primary vaccination
Population: The analysis was based on the Primary Total Vaccinated cohort, which included all vaccinated subjects with at least one vaccine dose documented.
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2963 | 520 | 520
Subjects | 1880 | 350 | 324

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 until 6 months following the last primary dose
Population: as for outcome 12
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2963 | 520 | 520
Subjects | 108 | 24 | 21

14. Secondary Outcome: Number of Subjects With AEs of Specific Interest (AESIs)
Description: An AESI was defined as an AE including autoimmune diseases and other mediated inflammatory disorders and assessed by the investigator as specific to the treatment administration.
Time Frame: From Day 0 until 6 months following the last primary dose or the receipt of the booster vaccination, whichever comes first
Population: as for outcome 12
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2963 | 520 | 520
Subjects | 108 | 22 | 15

15. Secondary Outcome: Number of Subjects With Seroresponse (90%) to Anti-PT, Anti-PRN and Anti-FHA
Description: Seroresponse (90%) was defined as the number of subjects showing a concentration above a threshold that leads to 90% seroresponse in the ActHIB group.
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 792 | 275 | 251
Subjects
  Anti-PT | 706 | 248 | 165
  Anti-PRN: number analyzed (Participants) | 789 | 275 | 250
  Anti-PRN | 741 | 250 | 194
  Anti-FHA: number analyzed (Participants) | 791 | 275 | 249
  Anti-FHA | 705 | 248 | 166

16. Secondary Outcome: Number of Subjects With Anti-PT, Anti-PRN and Anti-FHA Antibody Concentrations ≥ 5 EL.U/mL
Description: Seroresponse was defined as the number of subjects showing a concentration above a threshold that leads to 90% seroresponse in the ActHIB group.
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 792 | 275 | 251
Subjects
  Anti-PT | 789 | 275 | 249
  Anti-PRN: number analyzed (Participants) | 789 | 275 | 250
  Anti-PRN | 786 | 275 | 244
  Anti-FHA: number analyzed (Participants) | 791 | 275 | 249
  Anti-FHA | 791 | 275 | 249

17. Secondary Outcome: Number of Subjects With Anti-polyribosylribitol Phosphate (Anti-PRP) Antibody Concentrations ≥ 0.15 µg/mL and ≥ 1.0 µg/mL
Description: Evaluation of persistence of anti-PRP antibodies induced by three primary vaccine doses of Hiberix, and ActHIB, each co-administered with Pediarix, Prevnar 13 and Rotarix, or Pentacel co-administered with Engerix-B, Rotarix and Prevnar 13 prior to the booster dose of Hiberix, ActHIB or Pentacel at 15-18 months of age and evaluation of immunogenicity of a booster dose of Hiberix co-administered with Infanrix, ActHIB co-administered with Infanrix and Pentacel in terms of the percentage of subjects with anti-PRP concentrations ≥0.15 µg/mL, ≥1.0 µg/mL and GMCs one month after the booster dose.
Time Frame: Prior to the booster vaccination and 1 month after the booster vaccination
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 336 | 236 | 186
Subjects
  Anti-PRP ≥ 0.15 µg/mL; PRE vaccination: number analyzed (Participants) | 329 | 226 | 175
  Anti-PRP ≥ 0.15 µg/mL; PRE vaccination | 247 | 172 | 116
  Anti-PRP ≥ 0.15 µg/mL; POST vaccination | 336 | 235 | 186
  Anti-PRP ≥ 1 µg/mL; PRE vaccination: number analyzed (Participants) | 329 | 226 | 175
  Anti-PRP ≥ 1 µg/mL; PRE vaccination | 106 | 61 | 44
  Anti-PRP ≥ 1 µg/mL; POST vaccination | 333 | 231 | 184

18. Secondary Outcome: Anti-Hepatitis B (Anti-HBs) Antibody Concentrations
Description: Antibody concentrations were tabulated as geometric mean concentrations (GMCs) and expressedas milli-international units per milliliter (mIU/mL).
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 363 | 258 | 239
mIU/mL | 3684.3 [3287.0 to 4129.5] | 3545.6 [3067.8 to 4098.0] | 1573.4 [1302.6 to 1900.6]

19. Secondary Outcome: Number of Subjects With S.Pneumoniae Antibody Concentrations ≥ 0.05 µg/mL, ≥ 0.2 µg/mL and ≥1.0 µg/mL
Description: Evaluation of immunogenicity of a 3-dose primary vaccination course of Prevnar 13 co-administered with Hiberix, Rotarix and Pediarix, of Prevnar 13 co-administered with ActHIB, Rotarix and Pediarix and of Prevnar 13 co-administered with Pentacel, Rotarix and Engerix-B in terms of S.pneumoniae GMCs and antibody concentrations ≥ 0.05µg/mL, ≥ 0.2 µg/mL, ≥ 1.0 µg/mL at one month after the last dose of primary vaccination.
Time Frame: At 1 month after the last dose of primary vaccination
Population: The analysis was based on the Primary According-to-Protocol (ATP)cohort for immunogenicity, including all evaluable subjects with 3 vaccine doses administered and for whom assay results were available for antibodies against at least one antigen for the blood sample taken 1 month after the last vaccine dose.
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 389 | 270 | 247
Subjects
  ≥ 0.05 µg/mL, Anti-Pneumoniae 1: number analyzed (Participants) | 384 | 268 | 245
  ≥ 0.05 µg/mL, Anti-Pneumoniae 1 | 384 | 268 | 245
  ≥ 0.05 µg/mL, Anti-Pneumoniae 3: number analyzed (Participants) | 382 | 269 | 245
  ≥ 0.05 µg/mL, Anti-Pneumoniae 3 | 382 | 269 | 243
  ≥ 0.05 µg/mL, Anti-Pneumoniae 4: number analyzed (Participants) | 389 | 268 | 247
  ≥ 0.05 µg/mL, Anti-Pneumoniae 4 | 389 | 268 | 247
  ≥ 0.05 µg/mL, Anti-Pneumoniae 5: number analyzed (Participants) | 379 | 266 | 246
  ≥ 0.05 µg/mL, Anti-Pneumoniae 5 | 379 | 266 | 246
  ≥ 0.05 µg/mL, Anti-Pneumoniae 6A: number analyzed (Participants) | 381 | 267 | 244
  ≥ 0.05 µg/mL, Anti-Pneumoniae 6A | 381 | 267 | 244
  ≥ 0.05 µg/mL, Anti-Pneumoniae 6B: number analyzed (Participants) | 383 | 267 | 245
  ≥ 0.05 µg/mL, Anti-Pneumoniae 6B | 378 | 260 | 241
  ≥ 0.05 µg/mL, Anti-Pneumoniae 7F: number analyzed (Participants) | 386 | 269 | 246
  ≥ 0.05 µg/mL, Anti-Pneumoniae 7F | 386 | 269 | 246
  ≥ 0.05 µg/mL, Anti-Pneumoniae 9V: number analyzed (Participants) | 386 | 270 | 246
  ≥ 0.05 µg/mL, Anti-Pneumoniae 9V | 385 | 270 | 246
  ≥ 0.05 µg/mL, Anti-Pneumoniae 14: number analyzed (Participants) | 384 | 267 | 244
  ≥ 0.05 µg/mL, Anti-Pneumoniae 14 | 384 | 267 | 244
  ≥ 0.05 µg/mL, Anti-Pneumoniae 18C: number analyzed (Participants) | 380 | 267 | 244
  ≥ 0.05 µg/mL, Anti-Pneumoniae 18C | 380 | 267 | 244
  ≥ 0.05 µg/mL, Anti-Pneumoniae 19A: number analyzed (Participants) | 384 | 266 | 245
  ≥ 0.05 µg/mL, Anti-Pneumoniae 19A | 383 | 265 | 244
  ≥ 0.05 µg/mL, Anti-Pneumoniae 19F: number analyzed (Participants) | 384 | 268 | 245
  ≥ 0.05 µg/mL, Anti-Pneumoniae 19F | 384 | 268 | 245
  ≥ 0.05 µg/mL, Anti-Pneumoniae 23F: number analyzed (Participants) | 384 | 268 | 245
  ≥ 0.05 µg/mL, Anti-Pneumoniae 23F | 384 | 267 | 244
  ≥ 0.2 µg/mL, Anti-Pneumoniae 1: number analyzed (Participants) | 384 | 268 | 245
  ≥ 0.2 µg/mL, Anti-Pneumoniae 1 | 382 | 267 | 244
  ≥ 0.2 µg/mL, Anti-Pneumoniae 3: number analyzed (Participants) | 382 | 269 | 245
  ≥ 0.2 µg/mL, Anti-Pneumoniae 3 | 379 | 268 | 243
  ≥ 0.2 µg/mL, Anti-Pneumoniae 4: number analyzed (Participants) | 389 | 268 | 247
  ≥ 0.2 µg/mL, Anti-Pneumoniae 4 | 389 | 267 | 247
  ≥ 0.2 µg/mL, Anti-Pneumoniae 5: number analyzed (Participants) | 379 | 266 | 246
  ≥ 0.2 µg/mL, Anti-Pneumoniae 5 | 377 | 265 | 245
  ≥ 0.2 µg/mL, Anti-Pneumoniae 6A: number analyzed (Participants) | 381 | 267 | 244
  ≥ 0.2 µg/mL, Anti-Pneumoniae 6A | 379 | 265 | 243
  ≥ 0.2 µg/mL, Anti-Pneumoniae 6B: number analyzed (Participants) | 383 | 267 | 245
  ≥ 0.2 µg/mL, Anti-Pneumoniae 6B | 351 | 242 | 224
  ≥ 0.2 µg/mL, Anti-Pneumoniae 7F: number analyzed (Participants) | 386 | 269 | 246
  ≥ 0.2 µg/mL, Anti-Pneumoniae 7F | 386 | 269 | 246
  ≥ 0.2 µg/mL, Anti-Pneumoniae 9V: number analyzed (Participants) | 386 | 270 | 246
  ≥ 0.2 µg/mL, Anti-Pneumoniae 9V | 385 | 269 | 243
  ≥ 0.2 µg/mL, Anti-Pneumoniae 14: number analyzed (Participants) | 384 | 267 | 244
  ≥ 0.2 µg/mL, Anti-Pneumoniae 14 | 381 | 265 | 241
  ≥ 0.2 µg/mL, Anti-Pneumoniae 18C: number analyzed (Participants) | 380 | 267 | 244
  ≥ 0.2 µg/mL, Anti-Pneumoniae 18C | 377 | 267 | 244
  ≥ 0.2 µg/mL, Anti-Pneumoniae 19A: number analyzed (Participants) | 384 | 266 | 245
  ≥ 0.2 µg/mL, Anti-Pneumoniae 19A | 379 | 259 | 235
  ≥ 0.2 µg/mL, Anti-Pneumoniae 19F: number analyzed (Participants) | 384 | 268 | 245
  ≥ 0.2 µg/mL, Anti-Pneumoniae 19F | 383 | 267 | 244
  ≥ 0.2 µg/mL, Anti-Pneumoniae 23F: number analyzed (Participants) | 384 | 268 | 245
  ≥ 0.2 µg/mL, Anti-Pneumoniae 23F | 376 | 265 | 231
  ≥ 1.0 µg/mL, Anti-Pneumoniae 1: number analyzed (Participants) | 384 | 268 | 245
  ≥ 1.0 µg/mL, Anti-Pneumoniae 1 | 334 | 239 | 213
  ≥ 1.0 µg/mL, Anti-Pneumoniae 3: number analyzed (Participants) | 382 | 269 | 245
  ≥ 1.0 µg/mL, Anti-Pneumoniae 3 | 188 | 140 | 138
  ≥ 1.0 µg/mL, Anti-Pneumoniae 4: number analyzed (Participants) | 389 | 268 | 247
  ≥ 1.0 µg/mL, Anti-Pneumoniae 4 | 318 | 226 | 199
  ≥ 1.0 µg/mL, Anti-Pneumoniae 5: number analyzed (Participants) | 379 | 266 | 246
  ≥ 1.0 µg/mL, Anti-Pneumoniae 5 | 354 | 250 | 225
  ≥ 1.0 µg/mL, Anti-Pneumoniae 6A: number analyzed (Participants) | 381 | 267 | 244
  ≥ 1.0 µg/mL, Anti-Pneumoniae 6A | 357 | 253 | 229
  ≥ 1.0 µg/mL, Anti-Pneumoniae 6B: number analyzed (Participants) | 383 | 267 | 245
  ≥ 1.0 µg/mL, Anti-Pneumoniae 6B | 232 | 151 | 117
  ≥ 1.0 µg/mL, Anti-Pneumoniae 7F: number analyzed (Participants) | 386 | 269 | 246
  ≥ 1.0 µg/mL, Anti-Pneumoniae 7F | 379 | 264 | 239
  ≥ 1.0 µg/mL, Anti-Pneumoniae 9V: number analyzed (Participants) | 386 | 270 | 246
  ≥ 1.0 µg/mL, Anti-Pneumoniae 9V | 338 | 234 | 203
  ≥ 1.0 µg/mL, Anti-Pneumoniae 14: number analyzed (Participants) | 384 | 267 | 244
  ≥ 1.0 µg/mL, Anti-Pneumoniae 14 | 360 | 250 | 223
  ≥ 1.0 µg/mL, Anti-Pneumoniae 18C: number analyzed (Participants) | 380 | 267 | 244
  ≥ 1.0 µg/mL, Anti-Pneumoniae 18C | 361 | 256 | 229
  ≥ 1.0 µg/mL, Anti-Pneumoniae 19A: number analyzed (Participants) | 384 | 266 | 245
  ≥ 1.0 µg/mL, Anti-Pneumoniae 19A | 290 | 200 | 164
  ≥ 1.0 µg/mL, Anti-Pneumoniae 19F: number analyzed (Participants) | 384 | 268 | 245
  ≥ 1.0 µg/mL, Anti-Pneumoniae 19F | 357 | 254 | 231
  ≥ 1.0 µg/mL, Anti-Pneumoniae 23F: number analyzed (Participants) | 384 | 268 | 245
  ≥ 1.0 µg/mL, Anti-Pneumoniae 23F | 297 | 208 | 180

20. Secondary Outcome: Antibody Titers for Poliovirus Types 1, 2 and 3
Description: Antibody titers were given as geometric mean titers(GMTs).
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 478 | 334 | 331
Titers
  Anti-Polio 1: number analyzed (Participants) | 447 | 322 | 317
  Anti-Polio 1 | 570.8 [509.2 to 639.8] | 620.9 [540.1 to 713.7] | 136.0 [114.7 to 161.1]
  Anti-Polio 2 | 471.8 [416.7 to 534.1] | 389.9 [337.3 to 450.6] | 210.9 [181.9 to 244.5]
  Anti-Polio 3: number analyzed (Participants) | 456 | 323 | 311
  Anti-Polio 3 | 982.8 [870.1 to 1110.2] | 963.2 [843.7 to 1099.5] | 297.4 [253.3 to 349.1]

21. Secondary Outcome: Number of Subjects With Anti-HBs Antibody Concentrations Greater Than or Equal to Cut-off Values
Description: The cut-off values were defined as a concentration≥ 3.3 mIU/mL (seropositivity) and ≥ 10 mIU/mL (seroprotection).
Time Frame: At 1 month after last dose of primary vaccination
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 363 | 258 | 239
Subjects
  Anti-HBs≥ 3.3 mIU/ml | 362 | 257 | 239
  Anti-HBs≥ 10 mIU/ml | 362 | 257 | 239

22. Secondary Outcome: Anti-polyribosylribitol Phosphate (PRP) Antibody Concentrations
Description: as for outcome 3
Time Frame: Prior to the booster vaccination and 1 month after the booster vaccination
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 336 | 236 | 186
µg/mL
  PRE: number analyzed (Participants) | 329 | 226 | 175
  PRE | 0.498 [0.422 to 0.588] | 0.467 [0.385 to 0.567] | 0.380 [0.299 to 0.484]
  POST | 48.782 [42.000 to 56.659] | 40.293 [33.386 to 48.630] | 37.543 [30.535 to 46.158]

23. Secondary Outcome: Anti-Hepatitis B (Anti-HBs) Antibody Concentrations ≥10.0 mIU/mL and ≥6.2 mIU/mL
Description: Antibody concentrations were expressed as geometric mean concentrations (GMCs) and expressed as milli-international units per milliliter (mIU/mL).
Time Frame: Prior to the booster vaccination
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 316 | 207 | 167
mIU/mL | 268.3 [226.7 to 317.5] | 247.0 [199.8 to 305.3] | 156.4 [117.9 to 207.5]

24. Secondary Outcome: Number of Subjects With Anti-HB Antibody Concentrations ≥10.0 mlU/mL and ≥6.2mLU/mL
Description: The cut-off values were defined as a concentration≥ 6.2 mIU/mL (seropositivity) and ≥ 10 mIU/mL (seroprotection).
Time Frame: Prior to booster vaccination
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 316 | 207 | 167
Subjects
  Anti-HBs ≥ 6.2 mIU/mL | 311 | 199 | 156
  Anti-HBs ≥10.0 mIU/mL | 306 | 198 | 154

25. Secondary Outcome: Number of Subjects With Anti-PT, Anti-FHA and Anti-PRN Concentrations ≥ 5 EL.U/mL
Description: Evaluation of persistence of anti-PT, anti-FHA and anti-PRN antibodies induced by Pediarix or Pentacel and Engerix-B prior to the administration of a booster dose of Hib vaccine at 15-18 months of age and evaluation of immunogenicity of a booster dose of Infanrix co-administered with Hiberix, a booster dose of Infanrix co-administered with ActHIB and a booster dose of Pentacel with respect to anti-PT, anti-FHA and anti- PRN antibodies.
Time Frame: Prior to the booster vaccination and 1 month after the booster vaccination
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 336 | 235 | 186
Subjects
  Anti-FHA, PRE: number analyzed (Participants) | 329 | 225 | 174
  Anti-FHA, PRE | 328 | 223 | 171
  Anti-FHA, POST: number analyzed (Participants) | 335 | 235 | 185
  Anti-FHA, POST | 335 | 235 | 185
  Anti-PRN, PRE: number analyzed (Participants) | 327 | 225 | 177
  Anti-PRN, PRE | 279 | 174 | 130
  Anti-PRN, POST: number analyzed (Participants) | 332 | 234 | 186
  Anti-PRN, POST | 331 | 233 | 185
  Anti-PT, PRE: number analyzed (Participants) | 324 | 220 | 172
  Anti-PT, PRE | 243 | 168 | 81
  Anti-PT, POST | 335 | 235 | 186

26. Secondary Outcome: Anti-poliovirus Types 1, 2, and 3 Antibody Titres and Titres ≥ 8
Description: Antibody concentrations were tabulated as geometric mean titers (GMTs) and expressed as titers.
Time Frame: Prior to the booster vaccination
Population: The analysis was performed on the Booster ATP cohort for immunogenicity which included subjects for whom assay results were available for antibodies against at least 1 antigen for the blood sample taken 1 month after the administration of the booster vaccine dose.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 305 | 212 | 168
Titers
  Anti-polio 1: number analyzed (Participants) | 305 | 206 | 168
  Anti-polio 1 | 106.2 [91.1 to 123.8] | 101.6 [84.4 to 122.3] | 25.1 [20.3 to 31.0]
  Anti-polio 2: number analyzed (Participants) | 299 | 207 | 162
  Anti-polio 2 | 109.4 [92.8 to 129.1] | 89.5 [73.4 to 109.1] | 48.9 [39.7 to 60.2]
  Anti-polio 3: number analyzed (Participants) | 301 | 212 | 167
  Anti-polio 3 | 154.8 [129.3 to 185.3] | 151.9 [122.4 to 188.5] | 40.6 [31.4 to 52.5]

27. Secondary Outcome: Number of Subjects With Anti-Polio-1,2,3 Antibody Titers ≥ 8
Description: Anti-polio 1,2,3 antibody titers greater or equal to the cut off value were calculated.
Time Frame: Prior to booster vaccination
Population: as for outcome 26
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 305 | 212 | 168
Subjects
  Anti-polio 1 | 294 | 197 | 124
  Anti-polio 2 | 285 | 196 | 144
  Anti-polio 3 | 283 | 201 | 130

28. Secondary Outcome: Number of Subjects With Anti-D and Anti-T Antibody Concentrations ≥ 0.1 IU/mL and ≥1.0 IU/mL, Respectively.
Description: Evaluation of persistence of anti-D, anti-T antibodies induced by Pediarix or Pentacel and Engerix-B prior to the administration of a booster dose of Hib vaccine at 15-18 months of age and evaluation of immunogenicity of a booster dose of Infanrix co-administered with Hiberix, a booster dose of Infanrix co-administered with ActHIB and a booster dose of Pentacel with respect to anti-D and anti-T antibodies.
Time Frame: Prior to the booster vaccination and 1 month after the booster vaccination
Population: as for outcome 8
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 336 | 236 | 186
Subjects
  Anti-D≥ 0.1 IU/mL, PRE: number analyzed (Participants) | 329 | 226 | 177
  Anti-D≥ 0.1 IU/mL, PRE | 322 | 218 | 173
  Anti-D≥ 0.1 IU/mL, POST | 336 | 236 | 186
  Anti-T≥ 0.1 IU/mL, PRE: number analyzed (Participants) | 329 | 226 | 177
  Anti-T≥ 0.1 IU/mL, PRE | 292 | 196 | 154
  Anti-T≥ 0.1 IU/mL, POST | 336 | 236 | 186
  Anti-D≥1.0 IU/mL , PRE: number analyzed (Participants) | 329 | 226 | 177
  Anti-D≥1.0 IU/mL , PRE | 151 | 89 | 70
  Anti-D≥1.0 IU/mL , POST | 334 | 234 | 186
  Anti-T≥1.0 IU/mL , PRE: number analyzed (Participants) | 329 | 226 | 177
  Anti-T≥1.0 IU/mL , PRE | 52 | 27 | 14
  Anti-T≥1.0 IU/mL , POST | 330 | 233 | 180

29. Secondary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: as for outcome 10
Time Frame: Within 4 days (Days 0-3) following the booster dose
Population: Analysis was performed on the Booster Total Vaccinated cohort which included all subjects from Primary Total Vaccinated cohort that received the booster vaccine dose and had the symptom sheets completed.
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2224 | 416 | 379
Subjects
  Any Pain | 918 | 179 | 163
  Any Redness | 659 | 127 | 115
  Any Swelling | 392 | 82 | 75

30. Secondary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, fever and loss of appetite. Any = occurrence of any general symptom regardless of intensity grade or relationship to vaccination. Any fever= Axillary temperature equal to or above (≥) 38 degrees Celsius (°C).
Time Frame: Within 4 days (Days 0-3) following the booster dose
Population: as for outcome 29
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2225 | 416 | 379
Subjects
  Any Drowsiness | 857 | 164 | 119
  Any Irritability | 1293 | 250 | 201
  Any Loss of appetite | 614 | 141 | 85
  Any Fever | 119 | 18 | 20

31. Secondary Outcome: Number of Subjects With AEs of Specific Interest (AESIs)
Description: as for outcome 14
Time Frame: From booster dose until 6 months following receipt of the booster dose
Population: Analysis was performed on the Booster Total Vaccinated cohort which included all subjects from Primary Total Vaccinated cohort that received the booster vaccine dose.
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2337 | 435 | 400
Subjects | 47 | 12 | 7

32. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: as for outcome 12
Time Frame: Within 31 days (Day 0 to Day 30) following the booster dose
Population: as for outcome 31
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2337 | 435 | 400
Subjects | 882 | 159 | 138

33. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From the booster dose until 6 months following receipt of the booster dose
Population: as for outcome 31
Measure: Number; unit: Subjects
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 2337 | 435 | 400
Subjects | 29 | 4 | 2

34. Secondary Outcome: Anti-FHA, Anti-PRN and Anti-PT Antibody Concentrations
Description: as for outcome 4
Time Frame: pre-booster and one month after booster vaccination
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
Number analyzed (Participants) | 336 | 235 | 186
EL.U/mL
  Anti-FHA, PRE: number analyzed (Participants) | 329 | 225 | 174
  Anti-FHA, PRE | 41.3 [37.4 to 45.6] | 40.0 [35.2 to 45.5] | 22.7 [20.0 to 25.7]
  Anti-FHA, POST: number analyzed (Participants) | 335 | 235 | 185
  Anti-FHA, POST | 464.9 [430.0 to 502.7] | 492.5 [449.0 to 540.3] | 263.8 [239.5 to 290.5]
  Anti-PRN, PRE: number analyzed (Participants) | 327 | 225 | 177
  Anti-PRN, PRE | 13.3 [12.0 to 14.8] | 11.2 [9.8 to 12.9] | 9.7 [8.3 to 11.3]
  Anti-PRN, POST: number analyzed (Participants) | 332 | 234 | 186
  Anti-PRN, POST | 288.9 [260.4 to 320.5] | 259.2 [225.6 to 297.7] | 153.2 [128.5 to 182.6]
  Anti-PT, PRE: number analyzed (Participants) | 324 | 220 | 172
  Anti-PT, PRE | 8.5 [7.7 to 9.3] | 8.6 [7.7 to 9.7] | 4.8 [4.2 to 5.3]
  Anti-PT, POST | 90.9 [83.9 to 98.4] | 93.1 [84.1 to 103.1] | 75.3 [66.7 to 85.1]

ADVERSE EVENTS:
Time Frame: SAEs= Day 0 to 6 months following last primary dose and from booster dose until 6 months after receipt of booster dose. Systematically and non-systematically assessed frequent AEs=within 4 and 31 days following primary and booster vaccination respectively
Arm/Group | Hiberix Group | ActHIB Group | Pentacel Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 120/2963 | 24/520 | 21/520
Other Adverse Events (participants affected / at risk) | 2783/2963 | 495/520 | 488/520
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hiberix Group (N=2963) | ActHIB Group (N=520) | Pentacel Group (N=520)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cyanosis (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Cerebral palsy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Congenital aplastic anaemia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Congenital nystagmus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Congenital retinoblastoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Microcephaly (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Mitochondrial dna mutation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Developmental delay (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 16 (16) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Croup infectious (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Meningitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 10 (10) | 0 (0) | 2 (2)
Pertussis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 14 (14) | 2 (2) | 2 (2)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 13 (13) | 4 (4) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 9 (9) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 3 (3) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Child maltreatment syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (2)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 10 (10) | 3 (3) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Weight gain poor (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0)
Drooling (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dyskinesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 8 (8) | 3 (3) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Sympathomimetic effect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Autism spectrum disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Kawasaki's disease (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hiberix Group (N=2963) | ActHIB Group (N=520) | Pentacel Group (N=520)
Bronchiolitis (Infections and infestations) | 120 (123) | 20 (21) | 26 (26)
Conjunctivitis (Eye disorders) | 108 (114) | 29 (30) | 23 (25)
Cough (Respiratory, thoracic and mediastinal disorders) | 369 (427) | 64 (71) | 73 (89)
Decreased appetite (Metabolism and nutrition disorders) | 1596 (2761) | 304 (561) | 272 (460)
Diarrhoea (Gastrointestinal disorders) | 212 (231) | 36 (39) | 28 (34)
Erythema (Skin and subcutaneous tissue disorders) | 1306 (2465) | 262 (506) | 277 (525)
Irritability (Psychiatric disorders) | 2525 (6600) | 459 (1257) | 441 (1151)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 171 (195) | 33 (38) | 36 (41)
Otitis media (Infections and infestations) | 355 (420) | 63 (76) | 61 (79)
Pain (General disorders) | 2035 (4407) | 380 (906) | 383 (864)
Pyrexia (General disorders) | 1288 (1946) | 240 (360) | 201 (294)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 210 (241) | 45 (50) | 42 (45)
Somnolence (Nervous system disorders) | 2235 (5051) | 409 (960) | 387 (858)
Swelling (General disorders) | 944 (1547) | 191 (348) | 211 (370)
Teething (Gastrointestinal disorders) | 164 (204) | 30 (31) | 34 (41)
Upper respiratory tract infection (Infections and infestations) | 655 (787) | 109 (129) | 105 (124)
Vomiting (Gastrointestinal disorders) | 200 (231) | 36 (36) | 29 (31)

LIMITATIONS AND CAVEATS:
Anti-HBs antibody concentration cut off defining seropositivity was based on 6.2 mIU/mL instead of 3.3 mIU/mL for the pre-booster vaccination phase as tested by the commercial assay Centaur

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.